CLINICAL TRIAL: NCT02386475
Title: Effect of Serotonin and Levodopa Functional Recovery in Patients With Cerebral Infarction
Brief Title: Effect of Serotonin and Levodopa in Ischemic Stroke
Acronym: SELEIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SELEIS; 2014-000846-32 (EudraCT Number)
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups; Citalopram; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Interventions: Other: placebo
- citalopram 20 mg (Active Comparator): In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Interventions: Drug: citalopram
- sinemet plus 100 mg (Active Comparator): In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Interventions: Drug: sinemet plus
- Sinemet Plus + citalopram group (Active Comparator): In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Interventions: Drug: citalopram; Drug: sinemet plus

INTERVENTIONS:
Other: placebo — In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Other Names: control group
  Arms: Placebo
Drug: citalopram — In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Other Names: citalopram group
  Arms: Sinemet Plus + citalopram group; citalopram 20 mg
Drug: sinemet plus — In all cases, regardless of the assigned treatment group, will follow usual physiotherapy program and vascular risk factors, and treatment of stroke will be controlled according to current recommendations of the American Heart Association / American Stroke Association.
  Other Names: sinemet group
  Arms: Sinemet Plus + citalopram group; sinemet plus 100 mg

SUMMARY:
Cortical plasticity plays a pivotal role in functional recovery after a stroke. Neurotransmitter release, facilitates the creation of new synapses and promotes brain plasticity. In a pilot study, will evaluate the potential benefit of drugs that increase the release of neurotransmitters in patients with first stroke.

DETAILED DESCRIPTION:
Methods. Evaluate 240 consecutive patients with a first ischemic stroke with NIHSS 5-20 without aphasia and with a previous independent functional status (mRS <3). Patients will be randomized into four arms: 1) control group, 2) treatment with citalopram 20 mg / day, 3) group levodopa (sinemet plus)100 mg / day, 4) group levodopa (sinemet plus) 100 mg / day + citalopram 20 mg / day.

The treatment begins within the first 5 days of stroke and is maintained for 6 months. All patients will be treated according to current guidelines for secondary prevention. We will assess the following variables: demographic, vascular risk factors, etiologic subtypes according to TOAST criteria, neurologic deficit with the NIHSS scale, cognitive assessment with Minimental scale and functional status with scale modified Rankin at discharge, 3, 6 and 12 months, Symbol Digit Modalities Test (SDMT), GDS-15 Geriatric Depression Scale, Logical memory of WMS-IV . The cognitive assessment and motor functional status will be evaluated by a neuropsychologist and neurologist blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with a first stroke with NIHSS 5-20 points

  * Patients without aphasia to avoid interference in the assessment of depression and cognitive impairment
  * Patients with independent functional status prior to stroke (mRS <3)
  * Patients without prior cognitive impairment or depressive syndrome assessed by medical history with the patient and family.
  * The assigned treatment initiated within the first five days of stroke

Exclusion Criteria:

* • Patients with prior myocardial or cerebral hemorrhage

  * Patients with TIA
  * Patients with aphasia
  * History of cognitive impairment or prior depressive syndrome
  * Patients with no independent functional status mRS greater than or equal to 3
  * Underlying disease hopefully less than one year of life.
  * Patient pre-treatment with levodopa, an antidepressant or neuroleptic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Rankin Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Cocho, Principal Investigator — Hospital de Granollers
Locations (1):
- Granollers General Hospital, Granollers, Barcelnoa, Spain

REFERENCES:
- [Background] Thrift AG, Dewey HM, Macdonell RA, McNeil JJ, Donnan GA. Stroke incidence on the east coast of Australia: the North East Melbourne Stroke Incidence Study (NEMESIS). Stroke. 2000 Sep;31(9):2087-92. doi: 10.1161/01.str.31.9.2087. PMID 10978034
- [Background] Bruel-Jungerman E, Rampon C, Laroche S. Adult hippocampal neurogenesis, synaptic plasticity and memory: facts and hypotheses. Rev Neurosci. 2007;18(2):93-114. doi: 10.1515/revneuro.2007.18.2.93. PMID 17593874
- [Background] Jin K, Minami M, Lan JQ, Mao XO, Batteur S, Simon RP, Greenberg DA. Neurogenesis in dentate subgranular zone and rostral subventricular zone after focal cerebral ischemia in the rat. Proc Natl Acad Sci U S A. 2001 Apr 10;98(8):4710-5. doi: 10.1073/pnas.081011098. PMID 11296300
- [Background] Arvidsson A, Collin T, Kirik D, Kokaia Z, Lindvall O. Neuronal replacement from endogenous precursors in the adult brain after stroke. Nat Med. 2002 Sep;8(9):963-70. doi: 10.1038/nm747. Epub 2002 Aug 5. PMID 12161747
- [Background] Yamashita T, Ninomiya M, Hernandez Acosta P, Garcia-Verdugo JM, Sunabori T, Sakaguchi M, Adachi K, Kojima T, Hirota Y, Kawase T, Araki N, Abe K, Okano H, Sawamoto K. Subventricular zone-derived neuroblasts migrate and differentiate into mature neurons in the post-stroke adult striatum. J Neurosci. 2006 Jun 14;26(24):6627-36. doi: 10.1523/JNEUROSCI.0149-06.2006. PMID 16775151
- [Background] Sun Y, Jin K, Xie L, Childs J, Mao XO, Logvinova A, Greenberg DA. VEGF-induced neuroprotection, neurogenesis, and angiogenesis after focal cerebral ischemia. J Clin Invest. 2003 Jun;111(12):1843-51. doi: 10.1172/JCI17977. PMID 12813020
- [Background] Pariente J, Loubinoux I, Carel C, Albucher JF, Leger A, Manelfe C, Rascol O, Chollet F. Fluoxetine modulates motor performance and cerebral activation of patients recovering from stroke. Ann Neurol. 2001 Dec;50(6):718-29. doi: 10.1002/ana.1257. PMID 11761469
- [Background] Lim CM, Kim SW, Park JY, Kim C, Yoon SH, Lee JK. Fluoxetine affords robust neuroprotection in the postischemic brain via its anti-inflammatory effect. J Neurosci Res. 2009 Mar;87(4):1037-45. doi: 10.1002/jnr.21899. PMID 18855941
- [Background] Ruscher K, Kuric E, Wieloch T. Levodopa treatment improves functional recovery after experimental stroke. Stroke. 2012 Feb;43(2):507-13. doi: 10.1161/STROKEAHA.111.638767. Epub 2011 Nov 17. PMID 22096034
- [Background] Gu Q. Neuromodulatory transmitter systems in the cortex and their role in cortical plasticity. Neuroscience. 2002;111(4):815-35. doi: 10.1016/s0306-4522(02)00026-x. PMID 12031406
- [Background] Costa RM. Plastic corticostriatal circuits for action learning: what's dopamine got to do with it? Ann N Y Acad Sci. 2007 May;1104:172-91. doi: 10.1196/annals.1390.015. Epub 2007 Apr 13. PMID 17435119
- [Background] Jacobs BL, Fornal CA. Serotonin and motor activity. Curr Opin Neurobiol. 1997 Dec;7(6):820-5. doi: 10.1016/s0959-4388(97)80141-9. PMID 9464975
- [Background] Martinsson L, Hardemark H, Eksborg S. Amphetamines for improving recovery after stroke. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD002090. doi: 10.1002/14651858.CD002090.pub2. PMID 17253474
- [Background] Treig T, Werner C, Sachse M, Hesse S. No benefit from D-amphetamine when added to physiotherapy after stroke: a randomized, placebo-controlled study. Clin Rehabil. 2003 Sep;17(6):590-9. doi: 10.1191/0269215503cr653oa. PMID 12971703
- [Background] Platz T, Kim IH, Engel U, Pinkowski C, Eickhof C, Kutzner M. Amphetamine fails to facilitate motor performance and to enhance motor recovery among stroke patients with mild arm paresis: interim analysis and termination of a double blind, randomised, placebo-controlled trial. Restor Neurol Neurosci. 2005;23(5-6):271-80. PMID 16477089
- [Background] Gladstone DJ, Danells CJ, Armesto A, McIlroy WE, Staines WR, Graham SJ, Herrmann N, Szalai JP, Black SE; Subacute Therapy with Amphetamine and Rehabilitation for Stroke Study Investigators. Physiotherapy coupled with dextroamphetamine for rehabilitation after hemiparetic stroke: a randomized, double-blind, placebo-controlled trial. Stroke. 2006 Jan;37(1):179-85. doi: 10.1161/01.STR.0000195169.42447.78. Epub 2005 Dec 1. PMID 16322487
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] Petty GW, Brown RD Jr, Whisnant JP, Sicks JD, O'Fallon WM, Wiebers DO. Ischemic stroke subtypes : a population-based study of functional outcome, survival, and recurrence. Stroke. 2000 May;31(5):1062-8. doi: 10.1161/01.str.31.5.1062. PMID 10797166
- [Background] Grade C, Redford B, Chrostowski J, Toussaint L, Blackwell B. Methylphenidate in early poststroke recovery: a double-blind, placebo-controlled study. Arch Phys Med Rehabil. 1998 Sep;79(9):1047-50. doi: 10.1016/s0003-9993(98)90169-1. PMID 9749682
- [Background] Robinson RG, Schultz SK, Castillo C, Kopel T, Kosier JT, Newman RM, Curdue K, Petracca G, Starkstein SE. Nortriptyline versus fluoxetine in the treatment of depression and in short-term recovery after stroke: a placebo-controlled, double-blind study. Am J Psychiatry. 2000 Mar;157(3):351-9. doi: 10.1176/appi.ajp.157.3.351. PMID 10698809
- [Background] Bilge C, Kocer E, Kocer A, Turk Boru U. Depression and functional outcome after stroke: the effect of antidepressant therapy on functional recovery. Eur J Phys Rehabil Med. 2008 Mar;44(1):13-8. PMID 18385623
- [Background] Saxena SK, Ng TP, Koh G, Yong D, Fong NP. Is improvement in impaired cognition and depressive symptoms in post-stroke patients associated with recovery in activities of daily living? Acta Neurol Scand. 2007 May;115(5):339-46. doi: 10.1111/j.1600-0404.2006.00751.x. PMID 17489945
- [Background] Sonde L, Lokk J. Effects of amphetamine and/or L-dopa and physiotherapy after stroke - a blinded randomized study. Acta Neurol Scand. 2007 Jan;115(1):55-9. doi: 10.1111/j.1600-0404.2006.00728.x. PMID 17156266
- [Background] Dam M, Tonin P, De Boni A, Pizzolato G, Casson S, Ermani M, Freo U, Piron L, Battistin L. Effects of fluoxetine and maprotiline on functional recovery in poststroke hemiplegic patients undergoing rehabilitation therapy. Stroke. 1996 Jul;27(7):1211-4. doi: 10.1161/01.str.27.7.1211. PMID 8685930
- [Background] Yan T, Hui-Chan CW, Li LS. Functional electrical stimulation improves motor recovery of the lower extremity and walking ability of subjects with first acute stroke: a randomized placebo-controlled trial. Stroke. 2005 Jan;36(1):80-5. doi: 10.1161/01.STR.0000149623.24906.63. Epub 2004 Nov 29. PMID 15569875
- [Background] Cooke EV, Mares K, Clark A, Tallis RC, Pomeroy VM. The effects of increased dose of exercise-based therapies to enhance motor recovery after stroke: a systematic review and meta-analysis. BMC Med. 2010 Oct 13;8:60. doi: 10.1186/1741-7015-8-60. PMID 20942915